CLINICAL TRIAL: NCT02688140
Title: A Randomized Phase III Study to Compare Arsenic Trioxide (ATO) Combined to ATRA and Idarubicin Versus Standard ATRA and Anthracyclines-based Chemotherapy (AIDA Regimen) for Patients With Newly Diagnosed, High-risk Acute Promyelocytic Leukemia
Brief Title: Study for Patients With Newly Diagnosed, High-risk Acute Promyelocytic Leukemia
Acronym: TUD-APOLLO-064
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other); Groupe Francophone des Myelodysplasies (Other); HOVON - Dutch Haemato-Oncology Association (Other); Programa para el Tratamiento de Hemopatías Malignas (Unknown); German Federal Ministry of Education and Research (Other Government); Teva Pharmaceuticals Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-APOLLO-064
Record Dates: First submitted 2016-02-11; First posted 2016-02-23 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: APL; acute promyelocytic leukemia (M3); high-risk acute promyelocytic leukemia (APL/AML M3); acute myeloid leukemia with t(15;17)(q22;q12); newly diagnosed; high-risk
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Idarubicin; Cytarabine; Tretinoin; Mitoxantrone; Mercaptopurine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Induction therapy: Patients receive idarubicin i.v. over 20 minutes on day 1 and 3, oral tretinoin twice daily on day 1-28 (max. up to day 60) and arsenic trioxide i.v. over 2 hours on day 5-28 (max. up to day 60).
  In case of morphological CR and regenerated blood counts, consolidation therapy should be started within 2-4 weeks after documented CR.
  Consolidation therapy: Patients receive oral tretinoin twice daily on day 1-14. Treatment with tretinoin repeats every 4 weeks for up to 7 courses. Patients also receive arsenic trioxide i.v. over 2 hours on days 1-5 in week 1-4. Treatment with arsenic trioxide repeats every 8 weeks for up to 4 courses.
  Interventions: Drug: Arsenic trioxide; Drug: Idarubicin; Drug: Tretinoin
- Arm B (standard chemotherapy) (Active Comparator): Induction therapy: Patients receive idarubicin i.v. over 20 minutes on day 1,3,5 and 7, oral tretinoin twice daily on day 1-28 (max. up to day 60).
  In case of morphological CR and regenerated blood counts, consolidation therapy should be started within 2-4 weeks after documented CR.
  Consolidation I:
  IDA 5 mg/m2 i.v. day 1-4 Ara-C 1000 mg/m2/3h i.v. day 1-4 ATRA 45 mg/m2 p.o. day 1-15
  Consolidation II:
  MTZ 10 mg/m2 i.v. day 1-5 ATRA 45 mg/m2 p.o. day 1-15
  Consolidation III:
  IDA 12 mg/m2 i.v. day 1 Ara-C 150 mg/m2 every 8h i.v. day 1-5 ATRA 45 mg/m2 p.o. day 1-15
  Maintenance (duration 7 cycles = 2 years; one cycle lasts 106 days):
  6-MP 50 mg/m2 p.o. Cycle 1-7: day 1-91 (followed by 15 days of ATRA on days 92-106)
  MTX 15mg/m2 i.m./p.o. Cycle 1-7: once weekly for 91 days (followed by 15 days of ATRA on days 92-106)
  ATRA 45 mg/m2 p.o. Cycle 1-6: day 92-106 Cycle 7: without ATRA Administration
  (treatment break of 6-MP and MTX during ATRA administration)
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Tretinoin; Drug: Mitoxantrone; Drug: Mercaptopurine; Drug: Methotrexate

INTERVENTIONS:
Drug: Arsenic trioxide
  Other Names: ATO; Trisenox (R); As2O3
  Arms: Arm A
Drug: Idarubicin
  Other Names: IDA
Drug: Cytarabine
  Other Names: Ara-C
  Arms: Arm B (standard chemotherapy)
Drug: Tretinoin
  Other Names: all-trans retinoic acid; ATRA
Drug: Mitoxantrone
  Other Names: MTZ
  Arms: Arm B (standard chemotherapy)
Drug: Mercaptopurine
  Other Names: 6-Mercaptopurine; 6-MP
  Arms: Arm B (standard chemotherapy)
Drug: Methotrexate
  Other Names: MTX
  Arms: Arm B (standard chemotherapy)

SUMMARY:
Acute promyelocytic leukemia (APL) is a rare subtype of acute myeloid leukemia (AML) characterized by consistent clinical, morphologic, and genetic features. According to the FAB classification APL is designated as"M3 leukemia" and assigned to the WHO defined type of AML with recurrent cytogenetic abnormalities, "acute promyelocytic leukemia with t(15;17)(q22;q12), (PML/RARα) and variants".

Despite the dramatic progress achieved in frontline therapy of APL with ATRA plus anthracycline-based regimens, relapses still occur in approximately 20% of patients. Moreover, these regimens are associated with significant toxicities due to severe myelosuppression frequently associated with life-threatening infections and potentially serious late effects including development of secondary MDS/AML. In a recent randomized clinical trial in low/intermediate-risk APL (WBC ≤ 10 GPt/l APL0406 trial) a combination of arsenic trioxide (ATO) and ATRA has been shown to result into better survival with significantly lower toxicity rates compared to the standard ATRA + idarubicin (AIDA) therapy. Inspired by the results of this trial the investigators intend to perform a randomized study in high-risk APL (WBC at diagnosis > 10 GPt/l) comparing standard AIDA-based treatment with ATO/ATRA combination including low-doses idarubicin during induction. The investigators propose a modified ATO/ATRA protocol with the addition of two doses of IDA (50% compared to standard AIDA induction) for induction because of the anticipated need of adding anthracyclines to control hyperleukocytosis and to achieve long-term disease control in this high-risk APL population. This is followed by 4 cycles of ATO/ATRA consolidation therapy. As in the APL0406 study for low/intermediate-risk patients the investigators expect less severe hematologic toxicity and treatment-related mortality resulting in an improved outcome for patients in the experimental arm. Furthermore, from the start of consolidation, these patients (in contrast to the standard arm) can be treated on an outpatient basis, which is also considered to be associated with an improved quality of life. The study will be conducted as a European intergroup study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Women or men with a newly diagnosed APL by cytomorphology, confirmed by molecular analysis*
* Age ≥ 18 and ≤ 65 years
* ECOG performance status 0-3
* WBC at diagnosis > 10 GPt/l
* Serum total bilirubin ≤ 3.0 mg/dl (≤ 51 µmol/l)
* Serum creatinine ≤ 3.0 mg/dl (≤ 260 µmol/l)
* Women must fulfill at least one of the following criteria in order to be eligible for trial inclusion:
* Post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with Serum FSH > 40 U/ml)
* Postoperative (i.e. 6 weeks) after bilateral ovariectomy with or without hysterectomy
* Continuous and correct application of a contraception method with a Pearl Index of <1% (e.g. implants, depots, oral contraceptives, -intrauterine device - IUD)
* Sexual abstinence
* Vasectomy of the sexual partner

  * The confirmation of diagnosis at genetic level (microspeckled PML nuclear distribution by PGM3 monoclonal antibody and/or PML/RARa fusion by RT-PCR or fluorescence in situ hybridization (FISH) and/or demonstration of t(15;17) at karyotyping) will be mandatory for patient eligibility. However, in order to avoid delay in treatment initiation, patients can be randomized on the basis of morphologic diagnosis only and before the results of genetic tests are available

Exclusion Criteria:

* Patients who are not eligible for chemotherapy as per discretion of the treating physician
* APL secondary to previous radio- or chemotherapy for non-APL disease
* Other active malignancy at time of study entry (exception: basal-cell carcinoma)
* Lack of diagnostic confirmation at genetic level
* Significant arrhythmias, ECG abnormalities:
* Congenital long QT syndrome;
* History or presence of significant ventricular or atrial tachyarrhythmia;
* Clinically significant resting bradycardia (<50 beats per minute)
* QTc >500msec on screening ECG for both genders (using the QTcF formula detailed on protocol)
* Right bundle branch block plus left anterior hemiblock, bifascicular block
* Other cardiac contraindications for intensive chemotherapy (L-VEF <50%)
* Uncontrolled, life-threatening infections
* Severe non controlled pulmonary or cardiac disease
* Severe hepatic or renal dysfunction
* HIV and/or active hepatitis C infection
* Pregnant or breast-feeding patients
* Allergy to trial medication or excipients in study medication
* Substance abuse; medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results
* Use of other investigational drugs at the time of enrolment or within 30 days before study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-06; Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Event-free survival | From date of randomization until the date of first documented event, assessed up to 66 months
  events are: no achievement of haematological complete remission after induction therapy; no achievement of molecular remission after the last consolidation course; relapse; death including early death or development of secondary AML or MDS

SECONDARY OUTCOMES:
Rate of hematological complete remission | up to 60 days, from date of randomization until end of induction therapy
Rate of early death within 30 days after randomization | up to 30 days after randomization
Rate of overall survival (OS) | at 2 years
Rate of cumulative incidence of secondary MDS or AML | assessed up to 66 months, from date of randomization until occurance of secondary AML or MDS
Rate of cumulative incidence of relapse (CIR) | at 2 years
Incidence of hematological and non-hematological toxicity | assessed up to 30 months after randomization
Rate of molecular remission after the last consolidation cycle | up to 256 days after randomization
Assessment of acute promyelocytic leukemia/RARa transcript level reduction after induction therapy until end of study | assessed up to 30 months after randomization
Quality of Life at the end of induction therapy until the end of study | assessed up to 30 months after randomization
To investigate differences in the immune reconstitution between the two arms | assessed up to 30 months after randomization
Total hospitalization days during therapy | assessed up to 30 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof. Dr., Principal Investigator — Technische Universität Dresden (TUD)
Locations (8):
- French-Belgian-Swiss APL study group, Multiple Locations, France
- Germany (4):
  - AML-CG study group, Multiple Locations
  - AML-SG study group, Multiple Locations
  - OSHO study group, Multiple Locations
  - SAL study group, Multiple Locations
- GIMEMA study group, Multiple Locations, Italy
- HOVON study group, Multiple Locations, Netherlands
- PETHEMA study group, Multiple Locations, Spain

REFERENCES:
- [Derived] Platzbecker U, Ades L, Montesinos P, Ammatuna E, Fenaux P, Baldus C, Bernardi M, Berthon C, Bocchia M, Bonmati C, Borlenghi E, Bornhauser M, Carp D, Chantepie S, Crea E, Divona M, Dohner H, Ehninger G, Esteve Reyner J, Frayfer J, Garrido Diaz A, Gil C, Guarnera L, Hamm AF, Heiblig M, Heidenreich D, Kramer AJ, Ledoux MP, Lunghi M, Mancini V, Metzeler K, Miggiano MC, Muller-Tidow C, Peterlin P, Piciocchi A, Rieger K, Rollig C, Rossi G, Sanz MA, Serve H, Sohne M, Spiekermann K, Tavernier-Tardy E, Thiede C, Vives Polo S, Vogel W, Zappasodi P, Ziller-Walter P, Voso MT; SAL, AMCL-CG, AML-SG, OSHO, PETHEMA, HOVON and GIMEMA study groups. Arsenic Trioxide and All-Trans Retinoic Acid Combination Therapy for the Treatment of High-Risk Acute Promyelocytic Leukemia: Results From the APOLLO Trial. J Clin Oncol. 2025 Oct 10;43(29):3160-3169. doi: 10.1200/JCO-25-00535. Epub 2025 Aug 18. PMID 40825164